CLINICAL TRIAL: NCT05726968
Title: A Comparative Study on Three Different Doses of Intrathecal Hyperbaric Prilocaine With Fentanyl for Optimal Dose to be Used in Elderly Patients Undergoing Day Case Lower Abdominal and Urologic Surgeries.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Norhan Abdel Aleem Ali (Unknown); Hagar Hassanein Refaee (Unknown); Ahmed Abdullah Fathi Mohamed Almadawi (Unknown)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: MD-248-2022
Record Dates: First submitted 2022-11-16; First posted 2023-02-14 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2023-02

CONDITIONS: Three Different Doses of Intrathecal Hyperbaric Prilocaine With Fentanyl

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to determine the least sufficient dose of intrathecal hyperbaric prilocaine 2% combined with fentanyl 25 µg required for day-case lower abdominal and urologic surgeries , fewer adverse effects, faster recovery time, and shorter stay in post anesthesia care unit (PACU) in the geriatric patient population, as a previous study has investigated hyperbaric prilocaine (30 mg) when combined with fentanyl (20 µg) for a day-case perianal surgery, achieving a spinal anaesthesia with a mean sensory level of T9
Who Masked: Participant, Investigator
Masking Description: Patients will be randomly allocated to one of the 3 groups by sealed closed envelop technique
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ● Group P1 (N 15) (Active Comparator): Patients assigned to this group will receive intrathecal 30 mg (1.5 ml) of prilocaine 2% (Takipril, prilocaine hydrochloride 20 mg/mL, hyperbar, Sintetica) + 25 ug fentanyl (0.5 ml).
  Interventions: Drug: Pilocaine 2% (1.5 ml) and 25 ug fentany
- ● Group P2 (N 15) (Active Comparator): Patient assigned to this group will receive intrathecal 40 mg (2 ml) of prilocaine 2% + 25 ug fentanyl (0.5 ml).
  Interventions: Drug: Pilocaine 2% (1.5 ml) and 25 ug fentany
- ● Group P3 (N 15) (Active Comparator): patient assigned to this group will receive intrathecal 50 mg (2.5 ml) of prilocaine 2% + 25 ug fentanyl (0.5 ml)
  Interventions: Drug: Pilocaine 2% (1.5 ml) and 25 ug fentany

INTERVENTIONS:
Drug: Pilocaine 2% (1.5 ml) and 25 ug fentany — Patients will be randomly allocated into the study groups according to the list of random numbers. The study groups will be as follows:
  * Group P1 (N 15): patients assigned to this group will receive intrathecal 30 mg (1.5 ml) of prilocaine 2% (Takipril, prilocaine hydrochloride 20 mg/mL, hyperbar, Sintetica) + 25 ug fentanyl (0.5 ml).
  * Group P2 (N 15): patient assigned to this group will receive intrathecal 40 mg (2 ml) of prilocaine 2% + 25 ug fentanyl (0.5 ml).
  * Group P3 (N 15): patient assigned to this group will receive intrathecal 50 mg (2.5 ml) of prilocaine 2% + 25 ug fentanyl (0.5 ml).
  Other Names: Pilocaine 2%(2 ml) and 25 ug fentany; Pilocaine 2%(2.5 ml) and 25 ug fentany

SUMMARY:
To compare the effects of using different doses of intrathecal hyperbaric prilocaine 2% combined with fentanyl 25 µg in patients scheduled for a day-case lower abdominal and urologic surgery in the geriatric patient population.

DETAILED DESCRIPTION:
* To evaluate the safety and effectiveness of spinal anaesthesia with hyperbaric Prilocaine 2% in a reduced dose (30mg) in combination with Fentanyl (25µg) in day-case lower abdominal and urologic surgeries in the geriatric population.
* To compare between three different doses of prilocaine 2% in elderly patients undergoing day case lower abdominal and urologic surgeries.
* To estimate the duration of stay in PACU and hospital stay with different doses of prilocaine 2% in elderly patients undergoing day case lower abdominal and urologic surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age (65 - 80)
* ASA I - III
* Both genders.
* Height (1.60-1.90) m.
* BMI (18.5-40) kg m-2
* Scheduled for elective day-case lower abdominal or urologic procedures < 90 minutes in duration under spinal anesthesia.
* Type of surgery: Inguinal, femoral and incisional herniorrhaphies, bilateral varicocelectomies, hydrocelectomy, lymph node biopsies and mass excision biopsies, TURP surgery, Cystoscopies, ureteroscopy, bladder stone extraction, DJ insertion.

Exclusion Criteria:

* Patients requiring general anesthesia.
* Operations requiring sensory block above T10.
* Known or suspected coagulopathy (international normalised ratio > 1.4), thrombocytopenia (platelet count < 100,000).
* Known peripheral neuropathy, neurological deficits or skeletal deformities.
* Known allergy to prilocaine.
* Infection at site of injection.
* Patients' refusal to sign informed consent.
* Patients 'not meet inclusion criteria.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Duration of motor Block in hours | Through Study Completion,an average of 1day
  The primary outcome measure will be duration of motor Block in minutes, defined as the duration between intrathecal drug injection and time to unassisted ambulation or Bromage's score = 0 (no motor block).

SECONDARY OUTCOMES:
Onset of sensory block in minutes | Through Study Completion,an average of 1day
  Onset of sensory block, defined as the duration between intrathecal drug injection and complete absence of skin sensation to the pinprick test at T10 dermatome level in minutes.
Onset of motor block in minutes | Through Study Completion,an average of 1day
  Onset of motor block, defined as the duration between intrathecal drug injection and reaching a Bromage's score ≥ 2 in minutes.
Highest dermatomal level of sensory block. | Through Study Completion,an average of 1day
  Highest dermatomal level of sensory block.
Time to reach to highest sensory block in minutes. | Through study completion,an average of 1day
  Time to reach to highest sensory block in minutes.
Motor block at the time of reaching highest sensory block. | through study completion,an average of 1day
  Motor block at the time of reaching highest sensory block.
Full regression of sensory block | Through Study Completion,an average of 1day
  Full regression of sensory block, defined as the duration between intrathecal drug injection and regression to the S2 dermatome in minutes.
Duration of PACU stay | Through Study Completion,an average of 1day
  Duration of Post Anesthesia Care Unit stay in minutes.
The incidence of adverse effects | Through Study Completion,an average of 1day
  The incidence of adverse effects like hypotension, bradycardia, apnea, nausea, shivering, pruritus, block failure and pain during the operation. Failure to achieve a block level of T10 or additional analgesia request will be considered as block failure. Hypotension will be defined as a systolic blood pressure of < 90 mmHg or a decrease in mean arterial pressure of more than 20% from baseline preoperative value and bradycardia will be defined as heart rate < 50 beat/min.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Till Study Ending